CLINICAL TRIAL: NCT01024855
Title: Comparative Evaluation of Corneal Staining With Balafilcon A Lenses and Two Multi-Purpose Solutions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COBR-106-9608
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2012-03

CONDITIONS: Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RevitaLens OcuTec Multipurpose Solution (Investigational MPS) (Experimental)
  Interventions: Device: RevitaLens OcuTec MPS (Investigational MPS) and Opti-Free RepleniSH MPS (control)
- Opti-Free RepleniSH Multipurpose Solution (MPS, Control) (Active Comparator)
  Interventions: Device: RevitaLens OcuTec MPS (Investigational MPS) and Opti-Free RepleniSH MPS (control)

INTERVENTIONS:
Device: RevitaLens OcuTec MPS (Investigational MPS) and Opti-Free RepleniSH MPS (control) — multi-purpose lens care solution

SUMMARY:
A new multi-purpose solution (MPS)was clinically evaluated against Opti-Free RepleniSH MPS at specific time points over the course of four days. The study was conducted with PureVision lenses.

ELIGIBILITY:
Inclusion Criteria:

* were at least 18 years old;
* were experienced contact lens wearers;
* were correctable to at least 20/40 or better in both eyes with contact lenses;
* were in good general health, with healthy eyes (other than requiring vision correction);
* had not worn lenses for at least 12 hours before each baseline visit;
* had a corneal staining score no greater than Grade 1 in either eye at time of enrollment;
* had previously used an MPS or hydrogen peroxide solution successfully.

Exclusion Criteria:

* had a confirmed diagnosis of Sjögren's syndrome or other condition that results in a chronic and/or pathologic dry eye condition;
* required concurrent ocular medication or have used ocular medication within 24 hours of entering the study;
* had a known sensitivity or intolerance to any MPS, study products or ingredient(s);
* were currently participating in any other clinical study;
* had a condition or are in a situation that, in the investigator's opinion, may put them at significant risk, confound the study results, or interfere significantly with their participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott Medical Optics Inc., Santa Ana, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of employees occurred 7/8/2010 - 10/1/2010 thru employee bulletin for study taking place at in-house optometric clinic.
Pre-assignment Details: Prior to baseline visit subjects were instructed to undergo a "washout period" where no contacts were worn for 12 hours. Slit lamp exam was conducted prior to randomized group assignment. Eyes were thoroughly rinsed with unit-dose aline before pre-soaked study lenses were inserted.
Groups:
- RevitaLens and OptiFree: 30 subjects, one eye received RevitaLens MPS (investigational), one eye received Opti-Free RepleniSH MPS(control).
Period: Overall Study
Arm/Group | RevitaLens and OptiFree
Started | 30 (30 subjects enrolled in a paired/split-eye evaluation; each subject used both study treatments)
Completed | 29 (One subject of the 30 seen for baseline did not meet the inclusion/exclusion criteria)
Not Completed | 1
Not completed — Inclusion/exclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | RevitaLens and OptiFree
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants] — Study was performed in-house and strict confidentiality is required. Per Abbott In-House Study procedures, subject numbers and initials were used as identification. Limited access was given to data files to ensure confidentiality. Therefore, no gender data was collected for this study as it might reveal subjects identity to data entry personnel.
  participants
    Unknown | 30
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With No Change in Corneal Staining
Description: Subjects examined after corneal staining (a method used to assess the condition of the cornea) using a slit lamp to determine change from baseline and rated based on the following scale: 0=no change from baseline, 1=trace, 2=mild, 3=moderate, 4=severe.
Time Frame: Change from baseline after 1, 2, 4 and 6+ hours of wear
Population: per protocol
Measure: Number; unit: eyes
Groups:
- RevitaLens: 30 subjects, one eye received RevitaLens MPS (investigational).
- OptiFree: 30 subjects, one eye received Opti-Free RepleniSH MPS(control).
Arm/Group | RevitaLens | OptiFree
Number analyzed (Participants) | 30 | 30
eyes
  1 Hour - No Change | 16 | 17
  2 Hours - No Change | 19 | 14
  4 Hours - No Change | 21 | 21
  End of Day (>6 hrs) - No Change | 19 | 20

ADVERSE EVENTS:
Arm/Group | RevitaLens and OptiFree
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No